CLINICAL TRIAL: NCT05719480
Title: A Bidirectional Study in Exploring the Dynamic Changes of Plasma and Urine Metabolites During the Occurrence and Development of Liver Cancer in Southern China
Brief Title: A Bidirectional Study in Exploring the Dynamic Changes of Plasma and Urine Metabolites of Liver Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-441
Record Dates: First submitted 2022-12-21; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-12

CONDITIONS: Liver Cancer; Liver Cirrhosis; Fatty Liver; Hepatitis
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis; Fatty Liver; Hepatitis | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Liver Cancer patients: Patients who meet the diagnostic criteria of the Guidelines for Diagnosis and Treatment of Primary Liver Cancer (Version 2019) of the Chinese Medical Association
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- Liver Cirrhosis patients: Patients who meet the diagnostic criteria of the Guidelines for the Diagnosis and Treatment of Liver Cirrhosis (2019) issued by the Hepatology Branch of the Chinese Medical Association
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- Fatty Liver patients: Patients whose liver imaging findings meet the imaging diagnostic criteria for diffuse fatty liver disease or whose liver biopsy histology changes meet the pathological diagnostic criteria for fatty liver disease
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- Hepatitis patients: Patients who meet the diagnostic criteria for hepatitis B (ws 299-2008) and are diagnosed as hepatitis B;
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy
- healthy people: Healthy people without liver related medical history or other diseases known to affect blood lipid/protein metabolism
  Interventions: Diagnostic Test: Proteomics technology and liquid biopsy

INTERVENTIONS:
Diagnostic Test: Proteomics technology and liquid biopsy — using proteomics technology and liquid biopsy to investigate the changes of plasma and urine metabolites in different liver diseases during the development of liver cancer by collecting residual blood and urine from routine diagnosis and treatment or physical examination

SUMMARY:
The incidence of liver cancer in China shows a clear clinical path of hepatitis/fatty liver liver cirrhosis liver cancer. The dynamic changes of the internal environment on this pathway are important clues for early detection, diagnosis and even cure of liver cancer. The investigators carried out this study to investigate the changes of plasma and urine metabolites in different liver diseases during the occurrence and development of liver cancer.

DETAILED DESCRIPTION:
The process of liver cancer transformation is complex, so it is particularly important to explore the relationship between various liver diseases on its clinical pathway. Therefore, the investigators carried out this study to explore the changes of plasma and urine metabolites under different liver disease conditions during the development of liver cancer.

(1) Retrospective cohort: 600 patients were recruited, including 120 patients with hepatitis, 120 patients with cirrhosis, 120 patients with fatty liver, 120 patients with liver cancer, and 120 healthy people.,(2) Prospective cohort: 1400 patients were recruited, including 280 hepatitis patients, 280 cirrhosis patients, 280 fatty liver patients, 280 liver cancer patients, and 280 healthy people. During the course of the study, the subjects will not be given or provided with any randomized or any treatment driven by the study protocol. If it is clinically applicable, the treatment physician shall make the treatment decision and choose the treatment plan at his discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hepatitis B: patients who meet the WS299-2008 Diagnostic Standards for Hepatitis B issued by the Ministry of Health.
2. Patients with fatty liver: patients whose liver imaging findings meet the imaging diagnostic criteria for diffuse fatty liver disease or whose liver biopsy histology changes meet the pathological diagnostic criteria for fatty liver disease.
3. Patients with liver cirrhosis: patients who meet the diagnostic criteria of the Guidelines for the Diagnosis and Treatment of Liver Cirrhosis (2019) issued by the Hepatology Branch of the Chinese Medical Association;
4. Liver cancer patients: patients who comply with the Diagnostic and Treatment Standards for Primary Liver Cancer (2019 Edition) issued by the National Health Commission of the People's Republic of China.

Exclusion Criteria:

- 1. People who have a history of non research related liver diseases or other diseases known to affect blood metabolism (except for controlled type II diabetes); 2. Have a history of other malignant tumors, except for fully treated basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ; 3. Diseases requiring long-term use of immunosuppressive drugs (including steroids), including but not limited to congenital or acquired immunodeficiency diseases or active central nervous system metastatic cancer, active infection or uncontrolled heart disease; 4. Suffer from other uncontrolled serious diseases at the same time, such as unstable heart disease requiring treatment, diabetes with unsatisfactory control (fasting blood glucose>1.5 × Upper limit of normal value), mental illness and severe allergic history.

5. BMI is less than 18 or more than 25.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who met the diagnosis and criteria of hepatitis B,fatty live,liver cirrhosis or Liver cancer and were hospitalized in Southern Hospital of Southern Medical University.Subjects agreed to participate in the study and signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Achieve the expected number of enrolled cases | 3 years
  1. Retrospective cohort: 600 patients were recruited, including 120 patients with hepatitis, 120 patients with cirrhosis, 120 patients with fatty liver, 120 patients with liver cancer, and 120 healthy people.
  2. Prospective cohort: 1400 patients were recruited, including 280 hepatitis patients, 280 cirrhosis patients, 280 fatty liver patients, 280 liver cancer patients, and 280 healthy people.

CONTACTS AND LOCATIONS:
Overall Officials: jian guan, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China